CLINICAL TRIAL: NCT01333631
Title: Valproic Acid in Combination With Concurrent Chemoradiotherapy Using Gemcitabine for Unresectable Locally Advanced Pancreatic Cancer
Brief Title: Valproic Acid With Chemoradiotherapy for Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Dr. Konstantin lavrenkov, Soroka University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR513511CTIL
Record Dates: First submitted 2011-03-27; First posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-03

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced unresectable pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Valproic Acid

ARMS (1):
- Valporoic acid + chemoradiotherapy (Experimental)
  Interventions: Drug: Valproic acid

INTERVENTIONS:
Drug: Valproic acid — Valproic acid given concurrent with chemoradiotherapy for patients with pancreatic cancer

SUMMARY:
This is non-randomized phase 2 study to evaluate toxicity and efficacy of valproic acid (VA) with concurrent chemoradiotherapy (CCRT) containing weekly gemcitabine in patients with unresectable locally advanced pancreatic cancer (ULAPC). All patients will be planned for three-dimensional conformal radiotherapy (3-DCRT). A total dose of 54 Gy will be delivered using 2 Gy daily fractions given over 5 days a week.Intravenous (i.v.) chemotherapy (ChT) with gemcitabine 300 mg/m2 will be started at the first day of 3-DCRT.Total 5-6 weekly doses of i.v. ChT will be planned.VA will be administered orally in daily dose of 800 mg. Treatment with VA will be commenced at the first day and will be terminated at last day of RT.The patients will be followed till disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Newly-diagnosed, histologically/cytologically or CA 19.9 confirmed ULAPC
3. KPS > 60
4. No previous RT to abdomen
5. No serious comorbid condition Version 1, December 1, 2010
6. No treatment with biological response modifiers or cytotoxic agents within four weeks prior to study entry, apart from induction chemotherapy with gemcitabine
7. No participation in clinical trial using any investigational drug or device within four weeks prior to study entry
8. No serious complication of malignant condition
9. No previous or concurrent malignancy at other sites except cone biopsied in situ carcinoma of the uterine cervix and adequately treated basal cell or squamous cell carcinoma of the skin
10. Adequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

    * Hemoglobin > 9.0 Gm/dL
    * WBC count > 4.0x109/L
    * Neutrophile count > 1.5 cells x 109/L,
    * Platelet count > 100 x 109/L,
    * Creatinine < 1.5 mg/dL
    * Total bilirubin < upper limit of normal (ULN)
    * AST/SGOT < ULN
    * Calcium < ULN
11. Ability to sign informed consent
12. Ability to attend follow-up visits

Exclusion Criteria:

1. Operable disease
2. Distant metastases
3. KPS < 60
4. Previous RT to abdomen
5. Treatment with biological response modifiers or cytotoxic agents other then induction gemcitabine within four weeks prior to study entry
6. Participation in clinical trial using any investigational drug or device within four weeks prior to study entry
7. Major surgical procedure within two weeks prior to study entry
8. Serious comorbid condition, inclusive but not limited to myocardial infarction within previous six months, uncontrolled cardiac arrhythmias, uncontrolled angina pectoris, active infection including acute hepatitis
9. Serious complication of malignant condition
10. Previous or concurrent malignancy
11. Inadequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

    * Hemoglobin < 9.0 Gm/dL
    * WBC count < 4.0x109/L
    * Neutrophile count < 1.5 cells x 109/L,
    * Platelet count < 100 x 109/L,
    * Creatinine > 1.5 mg/dL
    * Total bilirubin > ULN (upper limit of normal)
    * AST/SGOT > ULN
    * Calcium > ULN
12. Inability to sign informed consent
13. Psychological, familial, sociological or geographical conditions which do permit regular medical follow-up and compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Number of the patients with side effects | 2 years

SECONDARY OUTCOMES:
Number of the patients survived | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Lavrenkov, MD, PhD, Principal Investigator — Soroka University Medical Center